CLINICAL TRIAL: NCT05378386
Title: Multicenter Post-Approval Study of Congenital Pulmonic Valve Dysfunction Studying the Edwards SAPIEN 3 Transcatheter Pulmonary Valve System With Alterra Adaptive Prestent
Brief Title: ALTERRA Post-Approval Study
Status: Active, not recruiting | Type: Observational
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-11
Record Dates: First submitted 2022-05-12; First posted 2022-05-18 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-07

CONDITIONS: Pulmonary Valve Insufficiency; Complex Congenital Heart Defect; Tetralogy of Fallot; Pulmonary Regurgitation; RVOT Anomaly
Keywords: Alterra prestent; SAPIEN 3; Pulmonic Delivery System; Transcatheter pulmonary valve replacement; Transcatheter pulmonary valve implantation
MeSH Terms: conditions — Pulmonary Valve Insufficiency; Tetralogy of Fallot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: Yes

GROUPS / COHORTS (1):
- TPVR: Transcatheter Pulmonary Valve Replacement
  Interventions: Device: Edwards Alterra Adaptive Prestent with SAPIEN 3 Transcatheter Pulmonary Valve System

INTERVENTIONS:
Device: Edwards Alterra Adaptive Prestent with SAPIEN 3 Transcatheter Pulmonary Valve System — The Edwards Alterra Adaptive Prestent is designed to reduce the diameter of large irregular right ventricular outflow tracts (RVOTs) and provide a circular, semi-rigid landing zone to place an Edwards SAPIEN 3 transcatheter heart valve (THV).

SUMMARY:
This study will monitor device performance and outcomes in subjects undergoing implantation of the Edwards SAPIEN 3 Transcatheter Pulmonary Valve System with Alterra Adaptive Prestent in the post-approval setting

DETAILED DESCRIPTION:
This is a single arm, prospective, multicenter post-approval study.

ELIGIBILITY:
Inclusion Criteria:

1. Native or surgically-repaired RVOT with severe PR
2. Clinically indicated for pulmonary valve replacement
3. Planned for treatment with the Alterra prestent and SAPIEN 3 THV

Exclusion Criteria:

1. Inability to tolerate an anticoagulation/antiplatelet regimen
2. Active bacterial endocarditis or other active infections

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with severe PR who have a native or surgically-repaired RVOT, are clinically indicated for pulmonary valve replacement, and are planned for treatment with the Alterra prestent and SAPIEN 3 THV
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-05-12 (Actual); Primary Completion 2025-09-25 (Actual); Study Completion 2035-07 (Estimated)

PRIMARY OUTCOMES:
Acute Device Success | 24 hours post-procedure
  Acute Device Success, defined as a non-hierarchical composite of:
  * Single Alterra deployed in the desired location
  * Single THV implanted in the desired location within Alterra
  * Right ventricle-pulmonary artery peak-to-peak gradient < 35 mmHg post-THV implantation
  * Less than moderate total pulmonary regurgitation (PR) by discharge transthoracic echocardiogram
  * Free of Alterra/SAPIEN 3 explant at 24 hours post-implantation

CONTACTS AND LOCATIONS:
Locations (24):
- United States (23):
  - Children's of Alabama, Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Cedars Sinai Medical Center, Los Angeles, California
  - Rady Children's Hospital, San Diego, California
  - Stanford University, Stanford, California
  - Colorado Children's Hospital, Aurora, Colorado
  - UF Health Shands Hospital, Gainesville, Florida
  - St. Joseph's Children's Hospital, Tampa, Florida
  - Advocate Children's Hospital, Oak Lawn, Illinois
  - Boston Children's Hospital, Boston, Massachusetts
  - Washington University in St. Louis, St Louis, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University, New York, New York
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Medical City Dallas, Dallas, Texas
  - Children's Memorial Hermann Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- Schneider Children's Medical Center of Israel, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No